CLINICAL TRIAL: NCT03316196
Title: Cognitive Training as a Novel Neuroscience-based Treatment for PTSD
Brief Title: Cognitive Training for PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MHBB-023-17S; CX001600-01A1 (Other Grant/Funding Number: VA)
Record Dates: First submitted 2017-10-10; First posted 2017-10-20 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Posttraumatic Stress Disorder
Keywords: trauma; PTSD; cognition
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Two arm randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- COGENT (Experimental): Participants will be Veterans assigned to the active cognitive training (see below for details).
  Interventions: Behavioral: COGENT COGNITIVE TRAINING
- Non-Training (Sham Comparator): Participants will be Veterans assigned to a non-training cognitive program matched for time and memory demands (see below for details).
  Interventions: Behavioral: Non training computer condition

INTERVENTIONS:
Behavioral: COGENT COGNITIVE TRAINING — Computer-administered cognitive training program. COGENT is a modified working memory capacity task designed to train cognitive functioning. COGENT was designed to contain high interference across trials. By requiring repeated practice with utilization of interference control across trials, COGENT is thought to enhance plasticity of cognitive systems and improve performance. That is, training is based on the premise that learning-based neural changes will occur via repeated exposure to a task demanding cognitive control resources
  Arms: COGENT
Behavioral: Non training computer condition — The non-training condition requires participants to complete a similar computer task for the same length of time. The non-training is a modified working memory capacity task designed to be inert. The non-training condition was designed to contain relatively less interference demands across trials. Participants are required to remember the same total number of items as in COGENT (i.e., storage requirements were equivalent), but the task contains relatively less interference inherent in the task.
  Arms: Non-Training

SUMMARY:
Posttraumatic stress disorder (PTSD) is a chronic, disabling condition that occurs in a subgroup of individuals after experiencing traumatic stress, and is common in Veterans seeking mental health treatment at the VA. Although evidence-based psychosocial treatments exist for PTSD, a substantial portion of individuals do not fully respond to treatment. Thus, there is a clear need to continue researching novel interventions for PTSD in Veterans. Recently, new interventions for mental health disorders have utilized computerized cognitive training techniques in order to improve the functioning of cognitive systems and reduce symptoms. This type of intervention, often referred to as neurotherapeutics, may hold promise for PTSD as a method for ameliorating symptoms and improving cognition. Individuals with PTSD demonstrate difficulties with cognitive control functions, which appear to be causally implicated in symptoms of the disorder (e.g., intrusive trauma-related memories). To date the efficacy of neurotherapeutics for PTSD has been understudied in Veterans.

The current proposal aims to bridge research on basic neurocognitive mechanisms of PTSD with intervention research by conducting a randomized controlled trial (RCT) of a cognitive control training program in 80 Veterans with PTSD. Veterans will complete computer-based training exercises designed to specifically target and improve aspects of cognitive control. Veterans will complete the program twice per week for eight weeks. Symptoms will be assessed before and after treatment, as well as at a two month follow up time point. The primary goal of the study is to examine the effect of the intervention on PTSD symptoms and cognitive deficits. Evaluating symptom change as a result of the intervention will provide critical data regarding the utility of this program as a PTSD treatment. If effective, this training program could serve as alternative treatment option for Veterans with PTSD, and could be translated into an easily transportable intervention for dissemination (e.g., through web-based platforms). A secondary goal is to use functional magnetic resonance imaging (fMRI) to better understand the mechanisms by which cognitive training culminates in symptom reduction. If training cognitive control with neurotherapeutics directly enhances functioning of specific neural substrates as hypothesized, improvements in affective processes relying on shared neural regions would also be predicted. Modifying functioning in these substrates with training may thus reduce symptoms by improving neural functioning while processing and managing trauma-related affect and information. Neural systems used for cognitive control targeted in the training described (e.g., dorsolateral prefrontal cortex [dlPFC]) are also recruited when individuals mentally manipulate emotional information, such as when individuals use reappraisal to change the way that they think about negative emotional situations or content. In this study, Veterans will complete a neutral cognitive control task and a reappraisal task while undergoing fMRI before and after completing the training treatment. This will be the first study to evaluate neurobiological mechanisms of this type of training in PTSD, which is a fundamental next step for understanding how to improve the training program and who may be best served by completing it.

DETAILED DESCRIPTION:
Posttraumatic Stress Disorder (PTSD) is one of the most prevalent service-related mental health conditions in treatment-seeking Veterans, yet even gold standard interventions are not universally effective. Veterans would be greatly served by development of novel intervention approaches for PTSD, particularly those could be easily transportable. The emerging field of neurotherapeutics, which uses computerized training techniques to modulate cognitive processing, is one such approach that has shown promise for improving cognitive and emotional symptoms in mental health disorders. The current proposal represents the first effectiveness study of a cognitive control training intervention for reducing PTSD symptoms in Veterans, with a goal of exploring neurobiological mechanisms of affective and cognitive generalization of training effects.

PTSD is characterized by deficits in "top-down" cognitive control abilities, as evidenced by neuropsychological findings of poor executive functioning and neurobiological evidence of diminished prefrontal cortical activity coupled with exaggerated limbic activity. Cognitive control deficits are causally implicated in re-experiencing symptoms, suggesting that cognitive control may be a novel and effective treatment target. The investigator developed a cognitive control training intervention that has demonstrated initial evidence of efficacy in civilian women with PTSD secondary to sexual assault. However, the effects of this program in Veteran participants and the precise neurocognitive mechanisms of symptom reduction in the intervention remain poorly understood. If training cognitive control directly enhances functioning of specific cognitive systems that are causally implicated in the etiology of emotional and cognitive symptoms, treatment-related improvements in affective symptoms and neuropsychological performance within the trained domain would be predicted. From a neurobiological perspective, training cognition is thought to operate via modification of specific neural substrates, suggesting that training effects should generalize to affective processes relying on shared neural regions. One such affective process is reappraisal (i.e., generating different ways of thinking about emotional content in order to regulate emotion), which requires cognitive control over affective emotional information, and depends on brain circuits identified as key cognitive control regions (e.g., dorsolateral prefrontal cortex, dlPFC). PTSD is characterized by aberrant affective and neurobiological patterns during reappraisal that likely contribute to persistent re-experiencing and hyperarousal symptoms. Training may reduce symptoms by improving neural functioning of cognitive control regions during affective control processes (e.g., reappraisal) that are critical to managing trauma-related affect.

In this proposal, the applicant's prior clinical trials research experience will be integrated with new mentoring in functional neuroimaging (fMRI) to facilitate identification of treatment-related symptom and neural change following cognitive control training. Bridging research on basic neurocognitive mechanisms of PTSD with intervention research in this way will ultimately facilitate precise neurotherapeutic treatment development and personalization techniques. In this randomized controlled trial (RCT), 80 Veterans with PTSD will be assigned to the cognitive control training program developed by the applicant (intervention condition: COGnitive ENhancement Training [COGENT]), or a minimal cognitive control program (sham training condition [ST]) completed twice week for 8 weeks. The COGENT training program requires participants to repeatedly utilize specific cognitive control functions (i.e., interference control) in the context of a modified working memory capacity task, with the goal of improving performance through implicit, practice-based learning. The primary outcome will be PTSD symptom reduction, and cognitive generalization will be assessed with a brief neuropsychological assessment. To evaluate changes in the neural bases proposed to underlie COGENT, participants will undergo fMRI while completing two cognitive control tasks (affectively neutral and emotionally balanced) before and after treatment. Assessments will occur at baseline, post-treatment, and at follow-up.

Aim 1: To examine the effects of the training program on PTSD and neurocognitive symptoms in Veterans. PTSD symptoms will be measured using the Clinician Administered PTSD Scale (CAPS) interview and neurocognitive functioning will be assessed with Delis Kaplan Executive Functioning System subtests. Individuals completing COGENT are hypothesized to show a) greater reduction in PTSD re-experiencing symptoms and b) improved neurocognitive performance relative to those in ST over time. Exploratory aims will also examine changes in PTSD diagnostic status across groups.

Aim 2: To examine neurobiological changes in COGENT versus ST during neutral and affective cognitive control tasks. Neurobiological response to treatment will be assessed using fMRI during cognitive control tasks (one affectively neutral working memory capacity task and one affectively balanced reappraisal task with negative emotional information). Individuals completing the COGENT program are predicted to demonstrate increased neural activation of dlPFC and anterior cingulate regions from pre- to post-training during the tasks. Exploratory aims will evaluate corresponding physiological change during the affective fMRI task and the utility of fMRI neural functioning at baseline for predicting treatment response.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants will be Veterans who:

* meet primary, current DSM-5 criteria for Posttraumatic Stress Disorder
* are literate in English
* intend to remain in the San Diego geographical area for the duration of the study
* are willing to attend assessment and treatment sessions

Exclusion Criteria:

* for the MRI portion, inability to safely complete fMRI session - unsafe metal in body, e.g.:

  * devices such as pacemakers
  * metal fragments in the skin like shrapnel
  * history of metal work or welding
  * history of eye surgery or washes because of metal
  * aortic/aneurysm clips
  * prosthesis
  * bypass surgery/coronary artery clips
  * hearing aids
  * heart-valve replacement
  * intrauterine devices with metal
  * shunts
  * electrodes
  * metal plates/pins/screws
  * neuro or bio-stimulators
  * older tattoos with metal ink
  * piercings the subject is unable or unwilling to remove
* uncorrectable vision problems
* claustrophobia
* inability to lie still on the back for approximately one hour
* inability to safely fit within the dimensions of the fMRI machine
* prior neurosurgery
* pregnancy or current breastfeeding (within 3 months)
* current IV drug use due to potential cerebrovascular effects
* or any other conditions that are deemed by Keck Imaging Center staff to contraindicated to safely complete the fMRI scanning
* a lifetime history of psychotic disorders
* lifetime history of bipolar disorder
* severe substance use disorder within the last year
* other psychiatric conditions that may adversely impact cognition and/or are deemed to require other primary psychological intervention
* history of any neurological disorder that might be associated with cognitive dysfunction, e.g.:

  * cerebrovascular accident
  * intracranial surgery
  * aneurysm
  * seizure disorder
* acute suicidality (defined as intent, plan, and/or attempt for severe self-harm within the past 3 months)
* or current circumstances that present a direct threat to the individual and require more imminent intervention, e.g.:

  * current domestic abuse
* individuals planning to begin medication changes within the time-frame of the study
* individuals currently undergoing evidence-based psychotherapy for PTSD
* individuals planning non-PTSD related psychosocial therapy change within the pre- to post-treatment time frame of the study
* those with life-threatening or acutely unstable medical conditions

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica A Bomyea, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | COGENT | Non-Training
Started | 42 | 39
Completed | 35 | 28
Not Completed | 7 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | COGENT | Non-Training | Total
Number analyzed (Participants) | 42 | 39 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.57 (8.53) | 37.77 (8.21) | 37.67 (8.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 29 | 24 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 12 | 29
  Not Hispanic or Latino | 25 | 27 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 0 | 5 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
  Black or African American | 3 | 4 | 7
  White | 29 | 20 | 49
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 7 | 3 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 39 | 81

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale - Reexperiencing
Description: This semi-structured interview is designed to measure posttraumatic stress disorder diagnostic status as well as symptoms severity. Total scores range from 0 to 20 with higher scores indicating greater severity; change over time will be evaluated.
Time Frame: Pre to Post Intervention (baseline to week 8)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COGENT | Non-Training
Number analyzed (Participants) | 35 | 28
score on a scale | 2.6 (2.9) | 2.96 (3.2)

2. Primary Outcome: Delis-Kaplan Executive Functioning System
Description: The Delis-Kaplan Executive Functioning System (DKEFS). This neuropsychological battery is designed to assess cognitive abilities in the executive functioning domain. Two relevant subtests, the Trail Making test and Color Word Interference Test, will be used. Total scores are calculated using a normed t score ranging from 0 to 100 with higher scores indicating better performance; change over time will be evaluated.
Time Frame: Pre to Post Intervention (baseline to week 8)
Population: Individuals who did not complete the neurocognitive assessment due to COVID protocols are not included in analyses
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COGENT | Non-Training
Number analyzed (Participants) | 18 | 12
score on a scale | -.36 (1.72) | -1.33 (1.19)

3. Secondary Outcome: Reading Span fMRI Task
Description: The Reading Span task is a working memory capacity assessment participants complete while undergoing functional MRI. Neural activation to task condition is measured using % signal change (0-100) with higher scores indicating greater activation; change over time will be evaluated.
Time Frame: Pre to Post Intervention (baseline to week 8)
Population: Individuals who did not complete the neurocognitive assessment due to COVID protocols are not included in analyses
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COGENT | Non-Training
Number analyzed (Participants) | 14 | 12
score on a scale | .47 (3.89) | 2.65 (2.22)

4. Secondary Outcome: Emotion Regulation fMRI Task
Description: The Emotion Regulation task is an assessment of how well participants can modulate their emotions in response to viewing images while undergoing functional MRI. Neural activation to task condition is measured using % signal change (0-100) with higher scores indicating greater activation; change over time will be evaluated.
Time Frame: Pre to Post Intervention (baseline to week 8)
Population: Individuals who did not complete the neurocognitive assessment due to COVID protocols are not included in analyses
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COGENT | Non-Training
Number analyzed (Participants) | 14 | 11
score on a scale | -.01 (.32) | .06 (.23)

5. Secondary Outcome: Clinician Administered PTSD Scale Diagnosis
Description: This semi-structured interview is designed to measure posttraumatic stress disorder diagnostic status as well as symptoms severity. Diagnostic status yes/no from the measure will be included as a secondary outcome (i.e., count of individuals with positive diagnosis).
Time Frame: Pre to Post Intervention (baseline to week 8)
Measure: Count of Participants; unit: Participants
Arm/Group | COGENT | Non-Training
Number analyzed (Participants) | 42 | 39
Participants | 21 | 16

ADVERSE EVENTS:
Time Frame: approximately 16 weeks
Arm/Group | COGENT | Non-Training
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/39
Other Adverse Events (participants affected / at risk) | 0/42 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-01-09): https://cdn.clinicaltrials.gov/large-docs/96/NCT03316196/Prot_000.pdf
  • Informed Consent Form (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/96/NCT03316196/ICF_001.pdf